CLINICAL TRIAL: NCT00247897
Title: What is the Best Skin Preparation Solution for Labour Epidural Analgesia? A Randomized Prospective Trial Comparing ChloraprepTM, DuraprepTM, and Chlorhexidine 0.5% in 70% Alcohol.
Brief Title: Comparing Skin Disinfectants Before Labour Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Roanne Preston, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: C05-0389
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Skin Bacteria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Skin antisepsis — See Detailed Description

SUMMARY:
The purpose of this study is to compare the current standard skin disinfectant solution for labour epidurals used at BC Women's Hospital to another common skin disinfectant and to the skin disinfectant solution recommended by the Public Health Agency of Canada (PHAC) prior to placing special intravenous lines. There is very little information available to guide doctors in deciding which is the best skin disinfectant for epidural analgesia. The study hypothesis is that the disinfectant solution recommended by the PHAC will be the most effective.

DETAILED DESCRIPTION:
Bacterial colonization of epidural catheters is known to occur and it has been suggested that catheter contamination occurs more frequently in the obstetric setting. Epidural catheters are usually colonized by the flora present at the skin insertion site and the rate of colonization varies from 5 to 30%. At present, there is a lack of scientific information available in order to make an evidence-based decision about skin disinfection prior to epidural analgesia. The labouring woman appears to have higher risk for infectious complications of epidural analgesia than other surgical patients.

All parturients considering a labour epidural who are admitted to Labour and Delivery at BC Women's Hospital during daytime weekday hours will be given an information sheet on the study by the Assessment room nurse. The Labour and Delivery Room nurses (which includes the Assessment room) are generally the first healthcare providers with whom women discuss labour epidural analgesia once admitted to hospital. All women interested in labour epidural analgesia who are admitted to Labour and Delivery, either via the Assessment room, or from one of the inpatient wards will be provided with the study information. After adequate time has been given for consideration of the study information, one of the researchers who is not directly involved in the patient's care will approach the patient for consent to participate in the study. This will happen prior to the actual request for labour epidural analgesia, therefore avoiding the point of pain at which the woman requires a labour epidural. Written consent will be obtained at that time. Upon request for a labour epidural, the woman will be randomized into one of 3 groups via a computer-generated randomization table (ZRandom). Group C will be ChloraprepTM, Group D: DuraprepTM, and Group S: chlorhexidine 0.5% in 70% alcohol.

Exclusion criteria include: temperature > 38oC orally at time of epidural request, local skin or generalized infection, systemic antibiotics administered prior to epidural request, presence of ruptured membranes > 24 hours, combined spinal-epidural analgesia planned, unable to speak/understand English, allergy to chlorhexidine or iodine, and patient refusal.

The attending anesthesiologist will wear a clean mask, clean his/her hands with either a wet scrub or alcohol-based antiseptic, and don sterile procedure gloves. Patients will be placed in either the left lateral, or sitting position according to anesthesiologist's preference. The skin overlying the lumbar interspaces will then be cleansed with the antiseptic solution, according to the recommended protocol for each solution.

Specific instructions for skin disinfection will be provided in an envelope to the attending anesthesiologist, according to the randomization group.

1. Subjects in the S group will have three applications of chlorhexidine 0.5% in 70% alcohol applied according to standard protocol. The chlorhexidine will be poured from a multi-use bottle into the sterile tray provided in the epidural kit. Sterile prep sponge sticks are part of the tray. Each sponge stick will be saturated with chlorhexidine and a 15 cm square area will be prepared over the L1-L5 interspaces using the centre-out method, allowing time for the solution to air-dry prior to proceeding.
2. Subjects in the D group will have their skin prepared with a single-use 6mL-unit applicator that contains a sterile, crushable ampoule of iodine 0.7% with 74% isopropyl alcohol. The solution is allowed to flow into the sponge tip via gravity and pumping action on the handle following activation of the applicator lever. A 15 cm square area over the L1-L5 interspaces will be covered using the centre-out method with a single application, and the solution will be allowed to air dry prior to proceeding.
3. Subjects in the C group will have their skin prepared with a single-use 10.5 mL-unit applicator that contains a sterile crushable ampoule of chlorhexidine gluconate 2% with isopropyl alcohol 70%. Following crushing the ampule with the outer wings of the sponge applicator, the solution will be pumped into the sponge tip until wet. A 15 cm square area over the L1-5 interspaces will be covered using the centre-out method with a single application. The solution will be allowed to air-dry prior to proceeding.

Epidurals will be placed between the L3 and L5 interspaces using a 17 gauge Tuohy needle, by loss of resistance to air or saline depending on operator choice. A 19 gauge Arrow flex tip endhole epidural catheter will be advanced to a depth of 4 to 6 cm within the epidural space. The catheter will be fixed in place by a sterile semi-permeable dressing (Tegaderm TM) and the proximal part of the catheter will be connected to a 0.2 micrometre filter. Standardized solutions of bupivacaine (0.08 or 0.125%) with fentanyl 2 micrograms/mL, prepared aseptically by the hospital pharmacy, will be used via the PCEA technique. Any initiation bolus, manual top-up, or top-up for surgical anesthesia will be prepared aseptically by the attending anesthesiologist as needed and injected into the epidural catheter through the filter.

There are no identifiable risks beyond potential reaction to the skin disinfectant. All of the skin preparation solutions are approved for skin disinfection prior to invasive/surgical procedures. There is no published data on the incidence of reaction to any of these products, and nothing that indicates one solution may have more inherent risk than the others.

Cultures and Microbiology

All skin culture samples will be taken by one of the researchers. All skin cultures will be obtained using sterile culture swabs (Copan Venturi Transport system) pre-moistened in sterile normal saline, taken from a 5 cm square area of skin. A baseline culture of skin flora at the proposed epidural insertion site will be taken prior to epidural insertion. The second culture will be taken immediately following skin antisepsis but before epidural insertion, to determine the initial efficacy of the antiseptic solution. The third culture will be taken following removal of the sterile occlusive dressing, immediately prior to epidural catheter removal. Prior to obtaining the epidural catheter tip for culture, the area of skin around the epidural catheter is disinfected with isopropyl alcohol. This is done to reduce the risk of skin contamination of the epidural catheter tip. Ten seconds later, the epidural catheter is removed by a researcher wearing a mask and sterile gloves, using sterile forceps, and the distal 3-4 cm is transacted with a sterile scissors.

The swabs will be coded, placed into 1.0 ml thioglycolate broth (BBL; Becton-Dickinson) and hand-delivered to the Microbiology lab at BC Children's and Women's Hospital. The tubes will then be spun for 1 minute to suspend organisms. Each swab and 0.1 ml aliquot of the suspension will then be inoculated onto blood agar plates. The epidural catheter tips will be placed in plain C+S containers and hand-delivered to the Microbiology lab where they will be rolled over blood agar plates. Standard culture techniques for the skin swabs and epidural catheter tips will be employed, to semi-quantitatively determine the bacterial count (colony-forming units or CFU's) and identify the micro-organisms. The CDC and PHAC definition for bacterial colonization of intravascular devices is a growth of 15 or more colony forming units/ml. We plan to use this as our definition for colonization of epidural catheters.

ELIGIBILITY:
Inclusion Criteria:

Request labour epidural analgesia. Able to understand English. No antibiotics taken in previous 24 hours. Membranes ruptured less than 24 hours. No current local or systemic infection. No contraindication to labour epidural analgesia

Exclusion Criteria:

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
25% reduction in skin bacterial colony counts at time of epidural catheter removal

SECONDARY OUTCOMES:
Skin bacterial colony count immediately following skin antisepsis. Bacterial growth on the epidural catheter tip at time of removal. Number of attempts at epidural insertion. Presence of blood in the epidural catheter at time of insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Roanne Preston, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital Labour and Delivery Suite, Vancouver, British Columbia, Canada